CLINICAL TRIAL: NCT00365131
Title: A Multicenter Study of the Efficacy of Cerezyme in Testing Skeletal Disease in Patients With Type I Gaucher Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC96-1101
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Gaucher Disease Type I; Cerebroside Lipidosis Syndrome; Clucocerebrosidase Deficiency Disease; Glucosylceramide Beta-Glucosidase Deficiency Disease; Gaucher Disease, Non-Neuronopathic Form
Keywords: Type I Gaucher disease; Glucocerebrosidase Deficiency Disease
MeSH Terms: conditions — Gaucher Disease | interventions — imiglucerase; Injections

INTERVENTIONS:
Drug: Cerezyme (imiglucerase for injection)

SUMMARY:
This is a multicenter, open-label, prospective study of the efficacy of Cerezyme in treating patients with skeletal manifestations secondary to Type I Gaucher disease.

The study objective is to evaluate and quantify skeletal responses as compared to baseline in Type I gaucher disease patients receiving Cerezyme therapy for 48 months. Additional objectives were to assess the usefulness of various skeletal parameters, such as bone pain, bone crises, bone mineral density, and serum and urine bone markers, as indicative of treatment response and may be useful in dose management.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Confirmed diagnosis of Type I Gaucher disease, with no prior enzyme replacement therapy, gene therapy or bone marrow transplantation, and who are ambulatory.
* Age 10-65 (patients 66-70 years of age are considered on a case-by-case basis following careful medical review).
* Dual energy X-ray absorptiometry (DEXA) of the femoral nech with a T-score ≤ -1.0.
* One of more of the following signs as documented by X-ray, computed tomography (CT), or magnetic resonance imaging (MRI), or symptoms of bone disease as documented in the patient's medical history or baseline examinations: a). history of at least one bone crises; b). Erlenmeyer flask deformity of the femora in children (10-17 years old); c). osteoarticular necrosis; d). medullary infarctions; e). lytic lesions; f). pathological fractures or fractures related to Gaucher disease; g). marrow infiltration to a degree such that Rosenthal's Magnetic Resonance Score was ≥ 3; h). bone density by quantitative computed tomography (QCT) or DEXA ≥ 1.5 standard deviation (SD) below age-adjusted normal value; and i). fat fraction ≤ 17%.

Exclusion Criteria:

* More than 1 joint replacement (revision surgery such as repair or replacement of a previously replaced joint is allowed).
* Pregnant, lactating or per-menopausal women.
* Active, uncontrolled infection, such as hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Major concurrent disorders (i.e. cancer, renal disease) or disorders known to affect bone (e.g. uncontrolled thyroid disease, hyperparathyroidism, hypoparathyroidism, gastrectomy, malabsorption, inflammatory bowel disease, rheumatoid arthritis, ankylosing spondylitis).
* Medications known to affect bone homeostasis (e.g. chronic oral corticosteroids, anticonvulsants, phenytoin and phenobarbital, hyper-physiological doses of estrogen, defined as > 0.625mg, or androgens, bisphosphates, calcitonin) within the first 2 months of the first Cerezyme infusion.
* Emotional, behavioral or psychological problems, which in the judgment of the principal investigator, would interfere with the patient adequately complying with the requirement of the study.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1997-12; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Skeletal response over 4 years of Cerezyme therapy
Assess use of skeletal parameter as indicative of treatment response and use in dose management

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Coral Springs, Florida, United States